CLINICAL TRIAL: NCT04390555
Title: COVID-19 in Hospitalised Patients With Preexisting CArdioVascular Diseases and/or Cardiac Involvement and/or Cardiovascular Risk Factors: the Global PCHF-COVICAV Registry
Brief Title: The Global PCHF-COVICAV Registry
Acronym: PCHF-COVICAV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: PCHF-COVICAV
Record Dates: First submitted 2020-05-06; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; Cardiovascular Diseases; Cardiovascular Risk Factor; Heart Failure
Keywords: COVID-19; Cardiovascular Diseases; Cardiovascular Risk Factor; Heart Failure
MeSH Terms: conditions — COVID-19; Cardiovascular Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CV involvement: Patients with COVID-19 and preexisting cardiovascular diseases and/or cardiovascular risk factors (diabetes mellitus, arterial hypertension and/or dyslipidaemia).
- Control: Patients with COVID-19 without preexisting cardiac involvement.

SUMMARY:
Background: Coronavirus disease (COVID-19) is a tremendous challenge the modern world has never seen before and is overwhelming the capacities of healthcare systems worldwide. Patients with cardiovascular diseases, heart failure in particular, and cardiovascular risk factors seem to be at a very high risk if affected by COVID-19 - and vice versa there are more and more reports of cardiac manifestations with the viral disease.

Aim: The purpose of the study is to characterise the clinical course of adult inpatients with COVID-19 and concomitant cardiovascular affection in a worldwide, multicentre PCHF registry.

Methods: Retrospective and prospective data analysis. Data on demographic, clinical, selected laboratory, electrocardiography and echocardiography parameters, treatment and outcome will be collected. The principal investigator provides dedicated electronic case report form. The primary outcome is in-hospital mortality. The secondary endpoints will be ICU length of stay, hospital length of stay, the need and duration of invasive mechanical ventilation, cardiovascular hospitalisation after 3 and 6 months from index hospitalisation, all-cause and cardiovascular mortality after 3 and 6 months from index hospitalisation.

ELIGIBILITY:
Inclusion Criteria:

* Adult inpatients (≥18 years old) with laboratory-confirmed COVID-19.

Exclusion Criteria:

* Age <18 years old.
* Outpatients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult inpatients (≥18 years old) with laboratory-confirmed COVID-19. Subjects with pre-existing cardiovascular disease and/or cardiac manifestations of COVID-19 infection (heart failure, acute coronary syndrome, myocarditis, arrhythmias, sudden cardiac arrest) and/or cardiovascular risk factors (dyslipidemia, hypertension, diabetes) are the focus of the study. Hospitalised subjects with COVID-19, but without cardiovascular disease or risk factors, will be used as a control population.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality. | Hospitalization period, assessed up to 30 days
  All-cause and cardiovascular mortality during index hospitalization.

SECONDARY OUTCOMES:
The length of stay in the intensive care unit. | Hospitalization period in the ICU, assessed up to 30 days
  The duration of hospitalization on the intensive care unit.
The duration of hospitalization. | Hospitalization period, assessed up to 30 days
  The total length of stay in the hospital.
The need and duration of invasive mechanical ventilation. | Hospitalization period, assessed up to 30 days
Hospitalization for cardiovascular causes or cardiovascular deaths within 3 months after hospitalization. | 3 months
Hospitalization for cardiovascular causes or cardiovascular deaths within 6 months after hospitalization. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Frank Ruschitzka, Prof. Dr. med, Study Director — University Hospital Zurich, Zurich, Switzerland; Andreas Flammer, PD Dr. med, Principal Investigator — University Hospital Zurich, Zurich, Switzerland; Mateusz Sokolski, MD, PhD, Principal Investigator — Wroclaw Medical University, Wroclaw, Poland
Locations (1):
- Zurich Heart Center, Unispital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruan Q, Yang K, Wang W, Jiang L, Song J. Clinical predictors of mortality due to COVID-19 based on an analysis of data of 150 patients from Wuhan, China. Intensive Care Med. 2020 May;46(5):846-848. doi: 10.1007/s00134-020-05991-x. Epub 2020 Mar 3. No abstract available. PMID 32125452
- [Background] Shi S, Qin M, Shen B, Cai Y, Liu T, Yang F, Gong W, Liu X, Liang J, Zhao Q, Huang H, Yang B, Huang C. Association of Cardiac Injury With Mortality in Hospitalized Patients With COVID-19 in Wuhan, China. JAMA Cardiol. 2020 Jul 1;5(7):802-810. doi: 10.1001/jamacardio.2020.0950. PMID 32211816
- [Background] Mehra MR, Desai SS, Kuy S, Henry TD, Patel AN. Cardiovascular Disease, Drug Therapy, and Mortality in Covid-19. N Engl J Med. 2020 Jun 18;382(25):e102. doi: 10.1056/NEJMoa2007621. Epub 2020 May 1. PMID 32356626 (Retraction: PMID 32501665 N Engl J Med. 2020 Jun 4;:)
- [Background] Cunningham JW, Ferreira JP, Deng H, Anker SD, Byra WM, Cleland JGF, Gheorghiade M, Lam CSP, La Police D, Mehra MR, Neaton JD, Spiro TE, van Veldhuisen DJ, Greenberg B, Zannad F. Natriuretic Peptide-Based Inclusion Criteria in a Heart Failure Clinical Trial: Insights From COMMANDER HF. JACC Heart Fail. 2020 May;8(5):359-368. doi: 10.1016/j.jchf.2019.12.009. Epub 2020 Mar 11. PMID 32171760
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Guo T, Fan Y, Chen M, Wu X, Zhang L, He T, Wang H, Wan J, Wang X, Lu Z. Cardiovascular Implications of Fatal Outcomes of Patients With Coronavirus Disease 2019 (COVID-19). JAMA Cardiol. 2020 Jul 1;5(7):811-818. doi: 10.1001/jamacardio.2020.1017. PMID 32219356
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Mehra MR, Ruschitzka F. COVID-19 Illness and Heart Failure: A Missing Link? JACC Heart Fail. 2020 Jun;8(6):512-514. doi: 10.1016/j.jchf.2020.03.004. Epub 2020 Apr 10. No abstract available. PMID 32360242
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Varga Z, Flammer AJ, Steiger P, Haberecker M, Andermatt R, Zinkernagel AS, Mehra MR, Schuepbach RA, Ruschitzka F, Moch H. Endothelial cell infection and endotheliitis in COVID-19. Lancet. 2020 May 2;395(10234):1417-1418. doi: 10.1016/S0140-6736(20)30937-5. Epub 2020 Apr 21. No abstract available. PMID 32325026